CLINICAL TRIAL: NCT02117908
Title: Application of CPAP to Reduce Complications and Improve Treatment of Radiofrequency Ablation of Lung Cancer Under Conscious Sedation. A Randomized Study
Brief Title: Study of the Application of CPAP to Reduce Complications and Improve Lung Cancer Ablation Radiofrequency Treatment
Acronym: CPAP-RFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Varea (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor-Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CPAP-RFP
Record Dates: First submitted 2014-04-11; First posted 2014-04-21 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-01

CONDITIONS: Atelectasis; Lung Cancer
Keywords: prevention; radiofrequency treatment; lung cancer ablation
MeSH Terms: conditions — Pulmonary Atelectasis; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP +4 cm H2O (Experimental): CPAP +4 cm H2O pressure using ResMedTM face mask
  Interventions: Device: RESMED AUTOSET S9
- ShamCPAP (Sham Comparator): shamCPAP using ResMedTM CPAP face mask modified for technical sham
  Interventions: Device: RESMED AUTOSET S9

INTERVENTIONS:
Device: RESMED AUTOSET S9 — Continuous positive pressure during surgery

SUMMARY:
The project aims to study whether the application of a continuous positive airway pressure (CPAP) of 4 cm water vapor is a safe method in pulmonary radiofrequency intervention (PRF) lung cancer under conscious sedation compared with placebo. And, assess whether CPAP prevents atelectasis formation and consequently reduces the potential complications of PRF and improves procedural success

ELIGIBILITY:
Inclusion Criteria:

* male and female aged 18 years and older
* Patient with a scheduled intervention for ablation of pulmonary malignant tumor with radiofrequency .
* Patient able to undergo tests and examinations required by the study.

Exclusion Criteria:

* Patients with CPAP intolerance test.
* Patients with progressive disease in which local treatment is not applicable
* Patients with intercurrent process (pleural effusion, pneumonia, ...).
* Patient unable to understand the proceedings.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | thirty days
  Patients with any of the following complications
  Pulmonary over-distention along intervention Pneumothorax along intervention Bronchial fistulas measures Computed tomography (CT)1, CT2 and CT3 Vomiting along intervention Decrease in MAP (mean arterial pressure) > 20% measured in the intraoperative period
  Assay of each of the previous complications

SECONDARY OUTCOMES:
Prevention of atelectasis. | during surgery
  Atelectasic area Normal ventilation pulmonary area Hypoventilation pulmonary area Hyperventilation pulmonary area Bronchial wall injury distance
Decrease associated complications with PFR. Measurement times: intraoperative, PACU (post-anesthesic care unit), hospital discharge, day 15 and day 30. | thirty days
  Major complications (death, failure to complete treatment, need for manual ventilation, intubation or resuscitation, pulmonary hemorrhage, need for pleural drainage, shock, fistulas, nerve injury, diaphragmatic injury, persistent pain, infections, increased hospitalization time and readmission rates) and any classified as a serious adverse event.
Treatment success | Measurement time: CT3
  Tumor ablation range, measured in CT3.
Predictors factors of the occurrence of complications during PRA (pulmonary radiofrequency ablation). | thirty days
  Minor complications (transient episodes of hypoxemia, apnea / hypoventilation or hypotension, pneumothorax without clinic symptoms or drainage, increased need for sedation, longer procedure) and any other event adverse not classified as serious.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique J Carrero Cardenal, MD PhD, Principal Investigator — Hospital Clínic i Provincial de Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Carrero-Cardenal E, Vollmer-Torrubiano I, Torres-Lopez M, Martin-Barrera G, Casanovas-Mateu G, Tercero-Machin FJ, Paez-Carpio A, Fabregas-Julia N, Valero-Castell R. Continuous positive airway pressure is unsafe for radiofrequency ablation of lung cancer under sedation: a randomised controlled trial. Insights Imaging. 2024 Jun 20;15(1):153. doi: 10.1186/s13244-024-01721-9. PMID 38900225